CLINICAL TRIAL: NCT01290874
Title: Blacks and Exacerbations on LABA vs. Tiotropium (BELT)
Brief Title: Blacks and Exacerbations on Long Acting Beta Agonists (LABA) vs. Tiotropium (BELT)
Acronym: BELT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Olmsted Medical Center (Other); American Academy of Family Physicians National Research Network (Network); Baim Institute for Clinical Research (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director of the Asthma Research Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010p001898
Record Dates: First submitted 2010-12-28; First posted 2011-02-07 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Asthma; Blacks; LABA; Tiotropium; Spiriva; African American; Serevent; salmeterol; Foradil; formoterol; Advair; Symbicort; Dulera
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tiotropium (Experimental): Tiotropium bromide will be evaluated as a treatment for asthma.
  Interventions: Drug: Tiotropium
- Salmeterol or Formoterol (Active Comparator): Long acting beta agonists (Serevent, Foradil) are the standard treatments for moderate asthma. The efficacy of Tiotropium will be compared to this standard.
  Interventions: Drug: Salmeterol; Drug: Formoterol

INTERVENTIONS:
Drug: Tiotropium — Tiotropium bromide 18 mcg once daily for one year of treatment.
  Other Names: Spiriva
  Arms: Tiotropium
Drug: Salmeterol — Salmeterol 50 mcg twice daily for one year of treatment.
  Other Names: Serevent
  Arms: Salmeterol or Formoterol
Drug: Formoterol — Formoterol 12 mcg twice daily for one year
  Other Names: Foradil
  Arms: Salmeterol or Formoterol

SUMMARY:
We are doing this study to learn how genes affect the way that people, specifically Black people, respond to treatment for asthma. Recent studies suggest that people respond differently to some asthma medications (eg Serevent, Foradil). Some people feel better when they use these inhalers, but others may not, and some people get worse. It seems that this difference shows up more often in Blacks than in Whites, which is why we are looking for Black subjects for this study. In all people, this difference seems to depend on their genes or DNA. This study is comparing the use of long acting asthma medications (Serevent, Foradil) to Tiotropium (Spiriva) for the treatment of asthma. Spiriva is used to treat chronic obstructive pulmonary disease (COPD). This study will help to see if this medication is also useful for treating asthma and whether it works better for some people than the current asthma medications.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disease that affects over 22 million people in the United States. Asthma produces 500,000 hospital admissions and accounts for 10.1 million days of lost work in adults annually. Asthma has been designated a priority condition of the Effective Health Care Program.

Blacks bear a disproportionate burden of asthma morbidity and mortality. In its 2005 report on ethnic disparities in health care, AHRQ identified hospital admissions for asthma as the second largest disparity in quality of health care for Blacks vs. Caucasians.

Long-acting beta-agonists (LABAs) produce extended increases in airway caliber among patients with asthma via action at the beta2-adrenergic receptor (ADRB2). Adding a LABA to an inhaled corticosteroid controller medication (ICS), can decrease asthma symptoms for many individuals and appears to decrease asthma exacerbations. LABA/ICS has become the most commonly prescribed ICS containing medication.

Drugs acting at ADRB2, including LABAs, have been associated with rare loss of long-term asthma control and increased serious adverse outcomes including death and respiratory failure, even when used with ICS. The risk appears four to five-fold greater in Blacks than non-Black patients with asthma.

Consensus guidelines recommend LABAs be added to ICS in those not completely controlled on ICS alone. These recommendations are based on weighing data on the benefit demonstrated in the general population vs. the rare risk of serious adverse outcomes and balancing the apparent benefits vs. the risks of LABAs (Kramer 2009). However, it appears that LABA/ICS may be significantly less effective in Blacks than Caucasians. Comparison of studies with LABA/ICS in Blacks vs. studies where Blacks were a small minority suggests that Blacks may have much less benefit than other racial groups. Additionally, recent data (Wechsler 2009) suggest that a polymorphism at the 16th position of the ADRB2 gene identifies a group of Blacks (those homozygous for arginine (Arg16Arg)) in whom the response of adding a LABA to an ICS is further diminished. This polymorphism is present in ~20% of US Blacks.

ELIGIBILITY:
Inclusion Criteria:

1. Black (self-identified, with at least one biological parent identified as Black)
2. Male and female subjects, ages 18-75
3. Ability to provide informed consent
4. Clinical history consistent with asthma for > 1 year.
5. Ability to perform pulmonary function tests
6. FEV1 > 40% of predicted
7. Receiving inhaled corticosteroids (ICS)/LABA combination therapy, or ICS moderate dose monotherapy and baseline ACQ>1.25
8. Non-smoker for past year (total lifetime smoking history < 10 pack-years)

Exclusion Criteria:

1. Use of greater than the equivalent of 1000 mcg inhaled fluticasone daily
2. Chronic use of oral corticosteroids or Anti IgE for asthma
3. Lung disease other than asthma or diagnosis of vocal cord dysfunction.
4. Significant medical illness (other than asthma) that is not stable.
5. Pregnancy or lactation or an unwillingness to maintain effective birth control.
6. History of a significant exacerbation of asthma or respiratory tract infection in the prior 4 weeks
7. History of life-threatening asthma requiring treatment with intubation and mechanical ventilation within 5 years.
8. Hypo sensitization therapy other than an established maintenance regimen.
9. Use of inhaled anticholinergic therapy (ipratropium, tiotropium) in prior month
10. Known contraindication to inhaled tiotropium e.g. narrow angle glaucoma, history of bladder neck obstruction or significant symptoms related to prostatic hypertrophy.
11. Inability to speak and read English.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2011-03-30; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (13):
- United States (13):
  - Edward Waters College Medical Center (Mayo), Jacksonville, Florida
  - Urban Family Practice, Marietta, Georgia
  - Albany Area Primary Healthcare, Inc, Newton, Georgia
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - G.A. Carmichael F.H.C., Canton, Mississippi
  - Swope Parkway Health Center, Kansas City, Missouri
  - UNYNET - Jefferson Family Medicine, Buffalo, New York
  - Montefiore Medical Group, The Bronx, New York
  - Carolinas Medical Center - NorthEast (Lovelace), Kannapolis, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Family Medicine Occupational Health Center, Shaker Heights, Ohio
  - BJHCHS - Hardeeville Medical Center, Ridgeland, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wechsler ME, Yawn BP, Fuhlbrigge AL, Pace WD, Pencina MJ, Doros G, Kazani S, Raby BA, Lanzillotti J, Madison S, Israel E; BELT Investigators. Anticholinergic vs Long-Acting beta-Agonist in Combination With Inhaled Corticosteroids in Black Adults With Asthma: The BELT Randomized Clinical Trial. JAMA. 2015 Oct 27;314(16):1720-30. doi: 10.1001/jama.2015.13277. PMID 26505596
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial enrollment began March 30, 2011 at the Asthma Research Center at Brigham and Women's Hospital. Subjects were recruited with print advertisements, internet postings, physician referrals, and by contacting patients in databases who asked to be contacted for studies.
Pre-assignment Details: Subjects on combination ICS/LABA were switched to equivalent-dose ICS monotherapy at the same time they were assigned to the Tiotropium vs. LABA arm of the study.
Period: Overall Study
Arm/Group | Tiotropium | Salmeterol or Formoterol
Started | 532 | 538
Completed | 122 | 134
Not Completed | 410 | 404

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Salmeterol or Formoterol | Total
Number analyzed (Participants) | 532 | 538 | 1070
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.6) | 45.1 (12.6) | 45.15 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 408 | 813
  Male | 127 | 130 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 36 | 67
  Not Hispanic or Latino | 501 | 502 | 1003
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 532 | 538 | 1070
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Asthma Exacerbation (Mean Number of Exacerbations/Person-year)
Description: We summarize the survival experience using mean number of exacerbations/person-year and compare it using the log-rank test comparing kaplan-meier survival curve.
Time Frame: evaluated monthly (on average) via questionnaire for 12 months
Population: intention-to-treat
Measure: Mean (95% Confidence Interval); unit: event per person-year
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 532 | 538
event per person-year | 0.37 [0.32 to 0.43] | 0.42 [0.36 to 0.48]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol or Formoterol; Test type: Superiority; p = 0.31, Log Rank

2. Secondary Outcome: Change in FEV1
Description: Average change in lung function (FEV1) evaluated by spirometry per participant over 12 months
Time Frame: from baseline to 12 months
Population: 255 and 253 participants are missing data on change in FEV1 in the Tiotropium and Salmeterol or Formoterol arms, respectively.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 277 | 285
liters | -0.018 [-0.047 to 0.012] | 0.003 [-0.026 to 0.031]

3. Secondary Outcome: Change in Asthma Control Questionnaire (ACQ)
Description: Average Change in Asthma Control Score Per Participant Over 12 Months Using the Asthma Control Questionnaire (ACQ).
  The ACQ has six questions regarding symptoms, rescue short-acting β-agonist use and one about FEV1 % predicted. A 7-point scale (0 = no impairment, 6 = maximum impairment) is used for each question and the ACQ score is the mean value of these questions - hence between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: from baseline to 12 months
Population: 334 and 326 participants are missing data on ACQ in the Tiotropium and Salmeterol or Formoterol arms, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 198 | 212
units on a scale | -0.70 [-0.81 to -0.60] | -0.66 [-0.77 to -0.55]

4. Secondary Outcome: Change in Asthma Quality of Life (AQLQ)
Description: Average Change in Asthma Quality of Life Score Per Participant Over 12 Months Using the Asthma Quality of Life Questionnaire (AQLQ).
  The AQLQ has 32 questions in four domains (symptoms, activity limitation, emotional function, and environmental stimuli) and measures the functional problems that are troublesome to individuals with asthma. Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items); 7-point Likert scale (7 = not impaired at all - 1 = severely impaired); scores range 1-7, with higher scores indicating better quality of life.
Time Frame: from baseline to 12 months
Population: 242 and 239 participants are missing data on AQLQ in the Tiotropium and Salmeterol or Formoterol arms, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 290 | 299
units on a scale | 1.00 [0.88 to 1.12] | 1.02 [0.90 to 1.14]

5. Secondary Outcome: Change in Asthma Symptom Utility Index (ASUI)
Description: Average Change in Asthma Symptom Utility Score Per Participant Over 12 Months Using the Asthma Symptom Utility Index (ASUI).
  The ASUI is an 11-item preference-based outcome measure used in clinical trials and cost-effectiveness studies for asthma and is designed to assess the frequency and severity of cough, wheeze, dyspnea, nighttime awakenings, and side effects, weighted according to patient preferences.
  4-point Likert scale to assess frequency (not at all, 1 to 3 days, 4 to 7 days, and 8 to 14 days) and severity (not applicable, mild, moderate and severe); scores range from 0 (worst possible symptoms) to 1 (no symptoms).
Time Frame: from baseline to 12 months
Population: 257 and 265 participants are missing data on ASUI in the Tiotropium and Salmeterol or Formoterol arms, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 275 | 273
units on a scale | 0.11 [0.09 to 0.13] | 0.10 [0.08 to 0.13]

6. Secondary Outcome: Change in Symptom-Free Day Questionnaire (SFDQ)
Description: Average Change in Symptom-Free Days Per Participant Over 12 Months Using the Symptom-Free Day Questionnaire (SFDQ).
  The asthma symptom free day questionnaire (SFDQ) quantifies the number of days with neither daytime nor nighttime asthma symptoms, nor awakenings due to asthma symptoms.
Time Frame: from baseline to 12 months
Population: The instrument used to collect data proved to be unreliable. The statistic for internal consistency demonstrated less than 30% internal consistency.
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Rescue Medication Use
Description: Average Change in Rescue Medication Use Per Participant Over 12 Months. Monthly questionnaires will evaluate the amount of rescue medication subjects have used on average, measured in puffs per day.
Time Frame: from baseline to 12 months
Population: 335 and 328 participants are missing data on rescue medication use in the Tiotropium and Salmeterol or Formoterol arms, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 197 | 210
units on a scale | -0.92 [-1.27 to -0.57] | -0.97 [-1.32 to -0.63]

8. Secondary Outcome: Change in Moderate Asthma Deterioration
Description: Average Change in Moderate Asthma Deterioration Per Participant Over 12 Months. The definition of a moderate asthma deterioration should include one or more of the following: deterioration in symptoms, deterioration in lung function, or increased rescue bronchodilator use. These features should last for 2 days or more, but not be severe enough to warrant systemic corticosteroid use and/or hospitalization.
Time Frame: from baseline to 12 months
Population: Inadequate baseline data was collected so that the change in this variable could not be assessed.
Arm/Group | Tiotropium | Salmeterol or Formoterol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of patient enrollment to up to 18 months after study completion.
Arm/Group | Tiotropium | Salmeterol or Formoterol
Serious Adverse Events (participants affected / at risk) | 84/532 | 69/538
Other Adverse Events (participants affected / at risk) | 338/532 | 342/538
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tiotropium (N=532) | Salmeterol or Formoterol (N=538)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Dysponea (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 8 (8) | 6 (6)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Localized Infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral cyst (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 23 (23)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tiotropium (N=532) | Salmeterol or Formoterol (N=538)
Disease Progression (General disorders) | 211 (211) | 203 (203)
Asthma (Respiratory, thoracic and mediastinal disorders) | 127 (127) | 139 (139)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No